CLINICAL TRIAL: NCT03573700
Title: SJCAR19: A Phase I/II Study Evaluating SJCAR19 (CD19-Specific CAR Engineered Autologous T-Cells) in Pediatric and Young Adult Patients ≤ 21 Years of Age With Relapsed or Refractory CD19+ Acute Lymphoblastic Leukemia
Brief Title: Evaluation of CD19-Specific CAR Engineered Autologous T-Cells for Treatment of Relapsed/Refractory CD19+ Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCAR19; NCI-2017-01399 (Registry Identifier: NCI Clinical Trial Registration Proogram)
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia, Refractory
Keywords: Leukemia; Leukemia, lymphoid; Leukemia, B-cell; Relapsed; Refractory; Pediatric; Chimeric antigen receptor; CAR; CAR T cell; Anti-CD19; CD19
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Lymphoid; Leukemia, B-Cell; Recurrence | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SJCAR19 Therapy (Experimental): Patients in both the Phase I and Phase II portion of the study will receive lymphodepleting chemotherapy (unless determined by PI that lymphodepletion is not necessary), followed by a single infusion of the patient-derived SJCAR19 cellular product. The most commonly used lymphodepleting chemotherapy regimen will consist of the agents: Fludarabine and Cyclophosphamide. They will also receive Mesna. Dosing of SJCAR19 on the Phase I study will follow a dose escalation schema, with dose changes based on dose-limiting toxicities. In the Phase II study, SJCAR19 dosing with follow the maximum tolerated dose, as determined in the Phase I portion.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Device: CliniMACS; Biological: CD19- specific CAR engineered autologous T-cells (SJCAR19 product)

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan
Drug: Fludarabine — Given IV
  Other Names: Fludara
Drug: Mesna — Given IV
  Other Names: Mesnex
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest.
Biological: CD19- specific CAR engineered autologous T-cells (SJCAR19 product) — Given IV

SUMMARY:
SJCAR19 is a research study seeking to evaluate the use of chimeric antigen receptor (CAR) T cell therapy, a type of cellular therapy, for the treatment of pediatric, adolescent and young adult patients with relapsed or refractory CD19+ acute lymphoblastic leukemia (ALL). CAR therapy combines two of the body's basic disease fighters: antibodies and T Cells. For this type of therapy, peripheral (circulating) immune cells are collected and then undergo a manufacturing process to engineer them to more effectively kill cancer cells. The SJCAR19 product will be manufactured at the St. Jude Children's Research Hospital's Good Manufacturing Practice (GMP) facility.

The main purpose of this study is to determine:

1. The largest dose of SJCAR19 that is safe to give,
2. How long SJCAR19 cells last in the body,
3. The side effects of SJCAR19, and
4. Whether or not treatment with SJCAR19 is effective in treating people with refractory or relapsed ALL.

DETAILED DESCRIPTION:
SJCAR19 is a Phase I/II clinical trial evaluating the use of SJCAR19 (CD19- specific CAR engineered autologous T-cells) in pediatric, adolescent and young adult patients with relapsed/ refractory CD19+ ALL. Treatment will include a single treatment course, with most patients receiving a lymphodepleting chemotherapy preparative regimen of fludarabine/ cyclophosphamide, followed by a single infusion of SJCAR19.

This protocol contains a 3-part consent process: 1) to proceed with autologous apheresis, 2) to proceed with manufacturing of the SJCAR19 product, and 3) to receive treatment with the SJCAR19 product (initially as Phase I, then proceeding to Phase II). The Phase I portion will evaluate the safety and maximum tolerated dose (MTD) of SJCAR19.

The Phase II portion will evaluate the efficacy, and provide further safety evaluation, of SJCAR19 in an expansion cohort at the MTD determined in the Phase I portion of the study. Additionally, for both the Phase I/II portions of the study there are correlative studies evaluating the biology of this treatment as well assessments into patient/caregiver experiences with undergoing this treatment.

ELIGIBILITY:
Inclusion Criteria for Autologous Apheresis:

* Age ≤ 21 years old
* CD19+ ALL with any of the following:

  * Minimal Residual Disease (MRD) ≥ 1% at end of up-front induction therapy
  * Hypodiploid (< 44 chromosomes or < 0.95 DNA index) CD19+ ALL with detectable disease at the end of up-front induction therapy
  * Increase in disease burden any time after the completion of up-front induction therapy
  * Primary refractory disease despite at least 2 cycles of an intensive chemotherapy regimen designed to induce remission
  * Refractory disease despite salvage therapy
  * 1st or greater relapse
* Estimated life expectancy of > 12 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥ 50
* Patients with a history of prior allogeneic hematopoietic cell transplantation [HCT] must be clinically recovered from prior HCT therapy, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to apheresis
* For females of child bearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment

Exclusion Criteria for Autologous Apheresis:

* Known primary immunodeficiency
* History of HIV infection
* Severe intercurrent bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products

Eligibility Criteria for Manufacturing SJCAR19:

* CD19+ ALL with any of the following:

  * Primary refractory disease despite at least 2 cycles of an intensive chemotherapy regimen designed to induce remission
  * Refractory disease despite salvage therapy
  * 2nd or greater relapse
  * Any relapse after allogeneic hematopoietic cell transplantation
  * 1st relapse if patient requires an allogeneic HCT as part of standard of care relapse therapy, but is found to be ineligible and/or unsuitable for HCT
* Age: ≤ 21 years of age
* Karnofsky or Lansky (age-dependent) performance score ≥ 50
* Estimated life expectancy of > 12 weeks
* Meets eligibility criteria to undergo autologous apheresis, or have previously undergone autologous apheresis

Inclusion Criteria for Treatment with SJCAR19:

* CD19+ ALL with any of the following:

  * Primary refractory disease despite at least 2 cycles of an intensive chemotherapy regimen designed to induce remission
  * Refractory disease despite salvage therapy
  * 2nd or greater relapse
  * Any relapse after allogeneic hematopoietic cell transplantation
  * 1st relapse if patient requires an allogeneic HCT as part of standard of care relapse therapy, but is found to be ineligible and/or unsuitable for HCT for any of the following reasons:

    * Patients that do not have an available allogeneic donor (defined as at least a 7/8 HLA-matched related/unrelated donor, 5/6 HLA-matched umbilical cord donor, or 3/6 HLA-matched haploidentical donor)
    * Patients with refractory leukemia, for which allogeneic transplant is known to be less effective in the B-ALL population, and
    * Patients who are unable to receive myeloablative total body irradiation (TBI), which is included in standard transplant regimens for patients with B - ALL.
* Detectable disease
* Age: ≤ 21 years of age
* Estimated life expectancy of > 8 weeks
* Prior to planned SJCAR19 infusion, patients with a history of prior allogeneic HCT must be at least 3 months from HCT, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to planned infusion
* Adequate cardiac function defined as left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%
* EKG without evidence of clinically significant arrhythmia
* Adequate renal function defined as creatinine clearance or radioisotope GFR ≥50 ml/min/1.73m2 (GFR ≥40 ml/min/1.73m2 if < 2 years of age)
* Adequate pulmonary function defined as forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing
* Karnofsky or Lansky (age-dependent) performance score ≥ 50
* Total Bilirubin ≤ 3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age
* Hemoglobin > 8 g/dl (can be transfused)
* Platelet count > 20,000/μL (can be transfused)
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For females of child bearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
  * If sexually active, agreement to use birth control until 6 months after T-cell infusion. Male partners should use a condom
* Available SJCAR19 product with ≥ 15% expression of the CD19-CAR, and killing of CD19+ targets ≥ 20% in an in vitro cytotoxicity assay
* Agreement to participate in long-term follow-up on protocol NCT00695279

Exclusion Criteria for Treatment with SJCAR19:

* CNS-3 disease with or without neurologic changes
* CNS-1/CNS-2 disease with neurologic changes
* Known primary immunodeficiency
* History of HIV infection
* Evidence of active, uncontrolled neurologic disease
* Severe, uncontrolled bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products
* Receiving systemic steroids therapy exceeding the equivalent of 0.5 mg/ kg/day of methylprednisolone, in the 7 days prior to CAR T-cell infusion
* Receiving systemic immunosuppressive therapy in the 14 days prior to CAR T-cell infusion
* Receiving intrathecal chemotherapy in the 7 days prior to CAR T-cell infusion

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee C. Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Talleur AC, Qudeimat A, Metais JY, Langfitt D, Mamcarz E, Crawford JC, Huang S, Cheng C, Hurley C, Madden R, Sharma A, Suliman A, Srinivasan A, Velasquez MP, Obeng EA, Willis C, Akel S, Karol SE, Inaba H, Bragg A, Zheng W, Zhou SM, Schell S, Tuggle-Brown M, Cullins D, Patil SL, Li Y, Thomas PG, Zebley C, Youngblood B, Pui CH, Lockey T, Geiger TL, Meagher MM, Triplett BM, Gottschalk S. Preferential expansion of CD8+ CD19-CAR T cells postinfusion and the role of disease burden on outcome in pediatric B-ALL. Blood Adv. 2022 Nov 8;6(21):5737-5749. doi: 10.1182/bloodadvances.2021006293. PMID 35446934
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was posted on http://clinicaltrials.gov. Potential patients were referred from their primary clinical service at St. Jude or through the Physician Referral Office and/or local providers. Twenty-four patients have been enrolled and started treatment since the study opened in July 2018.
Groups:
- Dose Escalation Level 1 (N = 6): Patients assigned to the first dose level of CD19 CAR T cells on the protocol dose escalation schema. Patients received lymphodepleting chemotherapy followed by a single infusion of 1x10^6 CAR+T cells /kg. Dose level changes were based on dose-limiting toxicities. See above 'Eligibility' for more details.
- Dose Escalation Level 2 (MTD) (N=18: Patients assigned to the second dose level of CD19 CAR T cells on the protocol dose escalation schema. Patients received lymphodepleting chemotherapy followed by a single infusion of 3x10^6 CAR+T cells /kg. Dose level changes were based on dose-limiting toxicities. See above 'Eligibility' for more details.
Period: Overall Study
Arm/Group | Dose Escalation Level 1 (N = 6) | Dose Escalation Level 2 (MTD) (N=18
Started | 6 | 18
Completed | 6 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Level 2 (MTD) (N=18): Patients assigned to the second dose level of CD19 CAR T cells on the protocol dose escalation schema. Patients received lymphodepleting chemotherapy followed by a single infusion of 3x10^6 CAR+T cells /kg. Dose level changes were based on dose-limiting toxicities. See above 'Eligibility' for more details.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Level 1 (N = 6) | Dose Escalation Level 2 (MTD) (N=18) | Total
Number analyzed (Participants) | 6 | 18 | 24
Age, Continuous [Median (Full Range); unit: years] | 11.2 [0.005 to 19.3] | 4.06 [0.44 to 17.9] | 6.07 [0.005 to 19.28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 15 | 20
  Black | 1 | 1 | 2
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose and Dose-limiting Toxicities
Description: The primary objectives for the Phase I study portion are to determine the maximum tolerated dose (MTD) and characterize the safety profile and dose-limiting toxicities (DLTs) of treatment with SJCAR19 in pediatric and young adult patient's ≤ 21 years of age, with relapsed or refractory CD19+ ALL. The proportion of participants with dose limiting toxicities are reported.
Time Frame: 4 weeks post-SJCAR19 infusion
Measure: Count of Participants; unit: Participants
Groups:
- Overall (N = 24): All patients treated on SJCAR19. See above 'Eligibility' for more details.
Arm/Group | Overall (N = 24) | Dose Escalation Level 1 (N = 6) | Dose Escalation Level 2 (MTD) (N=18)
Number analyzed (Participants) | 24 | 6 | 18
Participants | 2 | 1 | 1

2. Primary Outcome: Complete Response Rate
Description: The primary objective for the Phase II study portion is to evaluate the complete response (CR) rates of SJCAR19 in pediatric and young adult patient's ≤ 21 years of age, with relapsed or refractory CD19+ ALL.
Time Frame: 4 weeks post-SJCAR19 infusion
Measure: Count of Participants; unit: Participants
Groups:
- Overall (N = 24): All patients treated on SJCAR19.
Arm/Group | Overall (N = 24) | Dose Escalation Level 2 (MTD) (N=18) | Dose Escalation Level 1 (N = 6)
Number analyzed (Participants) | 24 | 18 | 6
Participants
  Response: Number of participants with Complete Response (MRD-positive or negative) status | 20 | 15 | 5
  Response: Number of patients with NR (No Response) | 4 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from on therapy up to 1 year post infusion.
Description: In the Phase I study, data on all adverse experiences/toxicities regardless of seriousness were collected. For Phase II (initial and any reinfusions), data on adverse events ≥ grade 3 were recorded. In addition, clinically significant grade 1-2 adverse events related/possibly related to the CAR T-cell product were collected.
Groups:
- Dose Level 1: Patients assigned to the first dose level of CD19 CAR T cells on the protocol dose escalation schema. Patients received lymphodepleting chemotherapy followed by a single infusion of 1x10^6 CAR+T cells /kg. Dose level changes were based on dose-limiting toxicities. See above 'Eligibility' for more details.
- Dose Level 2: Patients assigned to the second dose level of CD19 CAR T cells on the protocol dose escalation schema. Patients received lymphodepleting chemotherapy followed by a single infusion of 3x10^6 CAR+T cells /kg. Dose level changes were based on dose-limiting toxicities. See above 'Eligibility' for more details.
- Overall: All patients treated on SJCAR19. See above 'Eligibility' for more details.
Arm/Group | Dose Level 1 | Dose Level 2 | Overall
All-Cause Mortality (participants affected / at risk) | 3/6 | 9/18 | 12/24
Serious Adverse Events (participants affected / at risk) | 2/6 | 7/18 | 9/24
Other Adverse Events (participants affected / at risk) | 6/6 | 18/18 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=18) | Overall (N=24)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (3)
Fever (General disorders) | 0 (0) | 2 (2) | 2 (2)
Immune system disorders - Other (Immune system disorders) | 1 (1) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=18) | Overall (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (5) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 7 (7) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Apartate aminotransferase increased (Investigations) | 1 (1) | 5 (5) | 6 (6)
Blood bicarbonate decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 7 (7)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 8 (9) | 11 (12)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4) | 7 (9) | 9 (13)
Glucosuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 6 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 6 (6)
Hypertenison (Vascular disorders) | 0 (0) | 3 (3) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 8 (8) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 5 (5) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 4 (5) | 6 (7)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (4) | 9 (9) | 13 (13)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 10 (10)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 4 (4) | 7 (7) | 11 (11)
Pain in extremity (General disorders) | 2 (2) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 3 (3) | 7 (7) | 10 (10)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (4) | 2 (4)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
White blood cell decreased (Investigations) | 4 (4) | 10 (10) | 14 (14)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 8 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 5 (5) | 5 (5)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03573700/Prot_SAP_004.pdf
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03573700/ICF_005.pdf